CLINICAL TRIAL: NCT02214654
Title: A Pilot Study To Examine The Effects Of Ticagrelor To Protect Against Type 2 Diabetes-Induced Vascular Damage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Xiaofei Wang, Tianjin International Medical Center, Tianjin First Central Hospital
Other Study IDs: ISSBRIL0241
Record Dates: First submitted 2014-08-10; First posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes Mellitus；; Stable Coronary Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: None Retained — We will collect blood samples from the vena mediana cubiti, volume of sample blood will be 5ml.Centrifuge samples at 700gfor 20 min at 4 °C with no brake.Remove gently the upper phase (plasma) with a 5 ml pipette into a separate tube and store in 0.25 ml aliquots.Distribute 500 μl of samples into one isotype control and three sample tubes and add the special antibodies.Then account the CECs and sCD40/40L,etc.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ticagrelor，clopidogrel，antiplatelet drugs

SUMMARY:
The purpose of this study is to compare clopidogrel with ticagrelor which one has stronger anti-inflammation effect to protect against type 2 diabetes-induced vascular damage.

DETAILED DESCRIPTION:
i- Verify the study inclusion and exclusion criteria at visit 1.

ii- Inform patients (verbally and in writing) and their caregivers (when considered necessary and with the patient's consent) of the characteristics of the study and confirm their agreement to participate by signing the informed consent document.

iii- Assist with patient assessment, record the information in the case report form. Based on the data we get from the case report form, assign the patient to the experimental or control group by stratified randomization.

ⅳ- At visit 2 to obtain blood sample from peripheral vessel and analyze the density of CECs,sCD40L and hs-CRP by flow cytometry (FCM), ELISA and particle-enhanced turbidimetric immunoassay.

ⅴ- All patients are given aspirin 100mg/qd orally and the experimental group given ticagrelor 90mg/bid while the control group clopidogrel 75mg/qd for 30 days.

ⅵ- At visit 3 repeating step ⅳ and making comparison on numbers of CECs and CD40L between the two groups, and finish a statistic analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. A previous or new diagnosis of type 2 diabetes mellitus, document by one of following criteria:1）Hemoglobin A1c of ≥6.5% at diagnosis;2) Fasting plasma glucose (FPG) ≥126mg/dL (7.0 mmol/L);3) Two-hour plasma glucose≥200 mg/dL (11.1 mmol/L) during an oral glucose tolerance test (OGTT);4) with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose≥200mg/dL (11.1 mmol/L)( confirmed by repeat testing)
3. A previous or new diagnosis of stable CAD according to ICD 10 for at least 6 months, document by following criteria: 1) Stable angina; 2) No AMI or NSTE-ACS within 1 month;and(or) 3) EKG with ischemic ST-segment and(or) T-wave change; and(or)4) coronory artery stenosis ≥50% viewed by coronary CTA or coronary angiography
4. No medication history of clopidogrel/ticagrelor for at least 1 months
5. Female or male, and any race, aged≥18 years, not pregnant.

Exclusion Criteria:

1. Blood pressure>160/100 mm Hg;
2. Hypercholesterolemia(LDL-c >240mg/dl);
3. Hemoglobin A1c ≥ 10%;
4. Platelet count less than 10*10^9/L or hemoglobin <10 g/dL;
5. Intolerance or allergy to clopidogrel/ticagrelor or any of the excipients;
6. Patient with known inflammatory conditions or those on anti-inflammatory drug therapy;
7. Second and third degree atrioventricular block;
8. chronic obstructive lung disease or asthma;
9. Creatinine>2 mg/dl;
10. Malignancy;
11. Moderate or severe hepatic impairment;
12. History of intracranial haemorrhage;
13. Active pathological bleeding;
14. Pregnancy or lactation;
15. Any condition that increases the risk for noncompliance or being lost to follow-up;
16. Medicine history of potent CYP3A4 inhibitor(ketoconazole, clarithromycin,etc.);
17. No provision of informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be enrolled from outpatient and in hospital in Tianjin First Central Hospital
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
circulation endothelial cell | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofei Wang, doctor, Principal Investigator — Tianjin First Central Hospital
Locations (2):
- China (2):
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin